CLINICAL TRIAL: NCT07302178
Title: Effect of Combined Bitter Melon (Momordica Charantia L.) Extract and Snakehead Fish (Channa Striata) Powder Supplementation on Glycemic Status in Patients With Type 2 Diabetes Mellitus: A Randomized Controlled Trial
Brief Title: Combined Bitter Melon Extract and Snakehead Fish Powder Supplementation for Glycemic Control in Type 2 Diabetes
Acronym: BM-SF Glycemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Muhammadiyah Surakarta (Other)
Responsible Party: Principal Investigator, Fahrun Nur Rosyid, Head of Quality Assurance Group, Universitas Muhammadiyah Surakarta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMS-MOMORDICA-RCT2022
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Hyperglycemia
Keywords: Bitter melon extract; Momordica charantia; Channa striata; Glycemic status
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — bitter melon extract

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, parallel-group design evaluating the efficacy of a combined bitter melon extract and snakehead fish powder supplement compared with placebo for 4 weeks in adults with type 2 diabetes.
Masking Description: Both participants and study staff, including investigators and outcome assessors, will remain blinded to group allocation. The active supplement and placebo will be identical in appearance, packaging, and dosing schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of Snakehead Fish Powder + Bitter Melon Extract (Experimental): Participants in the experimental group will receive a combined herbal supplement containing Channa striata (snakehead fish) powder and Momordica charantia L. (bitter melon) extract.
  The supplement is provided in capsule form containing 500 mg per day, administered for 4 weeks.
  Interventions: Dietary Supplement: Snakehead Fish Powder + Bitter Melon Extract
- Placebo Capsule (Placebo Comparator): Participants in the control group will receive placebo capsules identical in appearance, administered once daily for 4 weeks, with no active herbal ingredients
  Interventions: Other: Placebo Capsule

INTERVENTIONS:
Dietary Supplement: Snakehead Fish Powder + Bitter Melon Extract — A 500 mg/day capsule containing a combination of:
  * Channa striata (snakehead fish) powder
  * Momordica charantia (bitter melon) ethanol extract Administered orally once daily for 4 weeks
  Arms: Combination of Snakehead Fish Powder + Bitter Melon Extract
Other: Placebo Capsule — Capsule identical in size, shape, and color to the intervention capsule, without active ingredients.
  Administered orally once daily for 4 weeks.
  Arms: Placebo Capsule

SUMMARY:
Type 2 diabetes mellitus (T2DM) remains a major global health problem due to its high prevalence, long-term complications, and substantial economic burden. Conventional antidiabetic therapies, including insulin and oral hypoglycemic agents, may cause significant side effects during long-term use and are contraindicated in certain clinical conditions. Therefore, safe and effective herbal-based alternatives are needed.

Previous preclinical and early clinical studies have shown that bitter melon (Momordica charantia L.) and snakehead fish (Channa striata) possess antidiabetic and anti-inflammatory properties, including improvement in glucose regulation, stimulation of insulin secretion, and regeneration of pancreatic cells. However, clinical evidence on their combined use remains limited.

This randomized, double-blind, placebo-controlled clinical trial aims to evaluate the effect of daily supplementation with a combination of bitter melon extract and snakehead fish powder on glycemic status in adults with Type 2 diabetes mellitus. Ninety eligible participants will be randomly assigned to a treatment group receiving 500 mg/day of the herbal combination or a placebo for 4 weeks. Glycemic status will be assessed primarily through glycated albumin (GA) levels.

The findings of this study are expected to provide scientific evidence regarding the safety and efficacy of this herbal combination as a complementary antidiabetic therapy.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a chronic metabolic disorder characterized by persistent hyperglycemia caused by impaired insulin sensitivity and progressive β-cell dysfunction. Long-standing hyperglycemia contributes to vascular inflammation, oxidative stress, and the formation of advanced glycation end products (AGEs), leading to complications that affect multiple organ systems including the kidneys, eyes, nerves, and cardiovascular system. The prevalence of T2DM continues to rise globally, particularly in low- and middle-income countries, resulting in a significant public health burden. Although conventional antidiabetic medications such as metformin, sulfonylureas, thiazolidinediones, and insulin effectively control blood glucose levels, long-term use may be associated with adverse effects including gastrointestinal disturbances, hypoglycemia, lactic acidosis, lipodystrophy, and contraindications in patients with hepatic or renal impairment. This situation highlights the need for safer, well-tolerated complementary approaches derived from natural products.

Bitter melon (Momordica charantia L.) has been traditionally used as a hypoglycemic agent and has demonstrated antidiabetic properties through multiple mechanisms, including reduction of glucagon secretion, inhibition of intestinal glucose absorption, enhancement of insulin release, and increased peripheral glucose uptake. Meanwhile, snakehead fish (Channa striata) is known to contain high levels of albumin, essential amino acids, and bioactive peptides that support tissue repair, modulate inflammation, and may contribute to improved pancreatic function. Preclinical studies and preliminary clinical observations suggest that these two natural ingredients possess synergistic potential in improving glycemic control, yet their combined effect has not been adequately evaluated in controlled human trials.

This study is designed as a randomized, double-blind, placebo-controlled clinical trial to assess the efficacy of a daily 500-mg supplementation of combined bitter melon extract and snakehead fish powder in improving glycemic status among adults with T2DM. A total of 90 eligible participants aged 20-65 years will be recruited from several community health centers in Surakarta, Indonesia. Participants will be randomized into intervention and placebo groups, while maintaining their standard antidiabetic therapy (metformin monotherapy). The intervention involves consuming one standardized capsule per day for four weeks. Bitter melon extract is prepared through ethanol maceration and evaporation, whereas snakehead fish powder is produced by steaming, drying, pulverizing, and sieving. Standardized nutrient and phytochemical analyses are conducted to ensure batch consistency and quality.

Glycemic control will be assessed primarily through measurements of glycated albumin (GA), which offers greater sensitivity to short-term glycemic fluctuations compared to HbA1c, and is particularly relevant for patients with variable glucose levels. Fasting plasma glucose will also be evaluated as a secondary outcome. Blood samples will be collected at baseline and at the end of week four. Statistical analyses will include paired t-tests for intragroup comparisons and independent t-tests for between-group comparisons, with significance set at p < 0.05.

This study is expected to generate scientific evidence on the efficacy and safety of the combined bitter melon-snakehead fish supplement as a complementary therapy for T2DM. The findings may contribute to the development of herbal-based antidiabetic products, support future patent applications, and provide a foundation for larger clinical trials aimed at improving accessible and culturally relevant diabetes management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes Mellitus (DMT2).
* Fasting plasma glucose ≥ 126 mg/dL and ≤ 200 mg/dL or random blood glucose between 200-300 mg/dL.
* Age 20-65 years
* Duration of diabetes 0-15 years.
* Currently using one class of oral antidiabetic medication (biguanide: metformin).
* Willing to participate and sign written informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding; or having impaired kidney or liver function (serum creatinine > 1.5 mg/dL; SGOT/SGPT > 2× upper limit).
* Allergy to snakehead fish powder (Channa striata) or bitter melon extract (Momordica charantia).
* Using antidiabetic medications other than metformin, or unable/unwilling to comply with study procedures.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Fasting Plasma Glucose (FPG) Level | Baseline and Week 4
  Fasting plasma glucose level measured at baseline (week 0) and after 4 weeks of supplementation with the combination of Channa striata (snakehead fish powder) and Momordica charantia (bitter melon extract), compared with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: FIK UMS, Principal Investigator — Universitas Muhammadiyah Surakarta

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves a limited sample size and contains sensitive clinical information. Data access is restricted to protect participant confidentiality and is limited to the research team as approved by the institutional ethics committee.